CLINICAL TRIAL: NCT02812745
Title: Is the Decrease in the Bispectral Index Correlated With a Decrease in Cardiac Output During the Induction of Anaesthesia? A Observational, Single-centre Study
Brief Title: Is the Decrease in the Bispectral Index Correlated With a Decrease in Cardiac Output During the Induction of Anaesthesia?
Acronym: BIS1
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI2015_843_0011
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Thoracic Surgery
Keywords: anaesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- patients: patients presenting an indication for general anaesthesia during elective cardiac surgery and being monitored for sedation depth
  * recording of cardiac output
  * other parameters
  Interventions: Device: recording of cardiac output; Device: other parameters

INTERVENTIONS:
Device: recording of cardiac output
Device: other parameters — BIS (bispectral index ), PI (perfusion index ), etCO2 (end-tidal carbon dioxide ), and brain NIRS (near-infrared spectroscopy)

SUMMARY:
Monitoring the bispectral index (BIS) as a peri-operative hemodynamic tool appears to be justified by the agreement between various clinical situations in which BIS monitoring appears to be of value: the prognosis in traumatic head injury, the diagnosis of brain death , and the diagnosis of amniotic fluid embolism. The current controversy concerning the "triple low" state reinforces the need for an accurate study in this field. Furthermore, the recent review by Bidd argues in this sense.

ELIGIBILITY:
Inclusion Criteria:

* Adult (over-18) patients presenting an indication for general anaesthesia during elective cardiac surgery and being monitored for sedation depth
* Good echogenicity
* Social security coverage

Exclusion Criteria:

* Pregnancy
* Subjects with black skin (a known technical limitation of plethysmography)
* Cardiac arrhythmia
* Sepsis
* Poor echogenicity
* Legal guardianship or incarceration
* Complications of anaesthesia during induction (anaphylactic shock, cardiac arrest, arrhythmia, or intubation not possible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting an indication for general anaesthesia during elective cardiac surgery and being monitored for sedation depth
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2015-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
correlation between variations in the BIS and variations in cardiac output | Day 0
  as measured by transthoracic echocardiography

SECONDARY OUTCOMES:
correlation between cardiac output and the perfusion index (PI) during the induction of anaesthesia. | Day 0
  measured by transthoracic echocardiography
correlation between cardiac output and end-tidal carbon dioxide (etCO2) during the induction of anaesthesia. | Day 0
  measured by transthoracic echocardiography
correlation between the cardiac output and the value of brain tissue oxygenation (measured by near-infrared spectroscopy (NIRS)) during the induction of anaesthesia | Day 0
  measured by transthoracic echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel LORNE, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France